CLINICAL TRIAL: NCT03967522
Title: CABRAMET: A Phase 2 Study of Cabozantinib in Metastatic Renal Cell Carcinoma (mRCC) With Brain Metastases
Brief Title: Evaluation of Cabozantinib in Metastatic Renal Cell Carcinoma (mRCC) With Brain Metastases
Acronym: CABRAMET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABRAMET (ET19-006)
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: mRCC; cabozantinib; brain metastases
MeSH Terms: conditions — Carcinoma, Renal Cell; Brain Neoplasms | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cabozantinib treatment (Experimental): All participants will be treated by 60 mg of cabozantinib once daily.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — All participants will be treated by 60 mg of cabozantinib once daily. Temporary or permanent discontinuation and/or dose reduction of cabozantinib therapy may be required for the management of some adverse reactions. When dose reduction is necessary, it is recommended to reduce to 40 mg daily, and then to 20 mg daily.

SUMMARY:
This is a multicenter, open-label, exploratory, single-arm, prospective phase II study to assess the efficacy and safety profile of cabozantinib in patients with brain metastases from metastatic renal cell carcinoma (mRCC).

DETAILED DESCRIPTION:
Cabozantinib is a small molecule inhibitor of tyrosine kinases which include MET (hepatocyte growth factor receptor protein), VEGFR (vascular endothelial growth factor receptors), AXL, RET (Rearranged during transfection), FLT3 (Fms-like tyrosine kinase-3), KIT (mast/stem cell factor receptor), ROS1, MER, TYRO3, TRKB (Tropomyosin receptor kinase B) and TIE-2 (angiopoietins receptor). Similar to other TKIs, cabozantinib is a reversible, ATP-competitive inhibitor. Cabozantinib has thus demonstrated significant activity in metastatic clear cell renal cell carcinoma after failure of one or 2 tyrosine kinase inhibitors and is now approved in the second line setting in Europe. Some efficacy was also demonstrated in patients in first line treatment when compared to sunitinib.

Brain metastasis in renal cancer are difficult to treat and cytotoxic systemic therapies are still not used, given by the more or less impermeable blood-brain barrier. The interest of cabozantinib in brain renal cell carcinoma metastases is encouraged by 3 recent cases reports of significant responses of brain metastases including a complete response of brain metastases in one case. Moreover MET receptor surexpression appear more frequent in brain metastases than in other renal cell carcinoma tumor sites. Cabozantinib as multitarget inhibitor including VEGF and MET receptors suggest that it could be a good option. Its efficacy in brain metastases from renal cell carcinoma requires further evaluation.

On this basis, the investigators propose to conduct an open-label exploratory single arm, multicenter prospective phase II trial to assess the efficacy of cabozantinib on brain metastases in metastatic renal cell carcinoma patients.

Ancillary studies:

The relationship between serum markers and efficacy data will be investigated. Serum and plasma sample will be collected at Baseline. MET expression and MET sequencing will be also performed on available tumor tissues.

ELIGIBILITY:
Inclusion Criteria:

I1. Age ≥ 18 years. I2. Histologically proven metastatic Renal Cell Carcinoma. I3. Brain metastases not requiring corticosteroids at dose > 40 mg/day. I4.At least 1 locally untreated brain lesion ≥8mm in longest diameter or >5mm if > 1 lesion.

I5.Not previously treated by cabozantinib. I6.Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) ≤ 1. I7.Life expectancy ≥ 3 months

I8.Adequate organ function as defined by the following criteria:

* Total serum bilirubin ≤ 2 x ULN (Gilbert's disease exempted)
* Serum transaminases and alkaline phosphatases ≤ 2.5 x ULN, or in case of liver or bone metastasis ≤ 5.0 x ULN
* Serum creatinine ≤ 2 x ULN OR creatinine clearance ≥ 50 ml/min
* Absolute neutrophil count (ANC) ≥ 1 500/mm3
* Platelets ≥ 100 000/mm3 (100 G/l)
* Hemoglobin ≥ 9.0 g/dl. I9. Covered by a medical/health insurance. I10. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

I11. Signed and dated IRB/ICE approved informed consent form. I12. Accepting to use effective contraception (barrier contraceptives) during study treatment and within at least 4 months after final dose of study therapy. Oral contraceptives are not acceptable.

Exclusion Criteria:

E1. Any local previous treatment of current brain metastases. E2. Any anti-coagulation therapy (except preventive treatment at low dose). E3. Contra-indication of Magnetic Resonance Imaging (MRI) (i.e. : pace-maker). E4. Uncontrolled seizures. E5. Any symptoms of intracranial hypertension. E6. Any of the following within 12 months prior to treatment initiation: severe/unstable angina, myocardial infarction, coronary artery bypass graft, symptomatic congestive heart failure, ischemic or hemorrhagic stroke including transient ischemic attack.

E7. Uncontrolled hypertension defined as systolic blood pressure >150 mmHg or diastolic pressure >90 mmHg, despite optimal medical treatment.

E8. Ongoing cardiac dysrhythmia of grade ≥ 2, atrial fibrillation of any grade, QTc interval > 0.43.

E9. Pregnant or breast feeding woman (mandatory negative serum or urinary pregnancy test at study entry for all women of childbearing potential).

E10. Any acute or chronic medical or psychiatric condition or laboratory abnormality that would make the patient unsuited to study participation.

E11. Any second malignancy within the last 3 years with the exception of basal cell carcinoma, in situ cervical cancer and pT1/a bladder cancer with no evidence of recurrent disease for 12 months.

E12. Patients receiving strong inhibitor or inducer of CYP3A4 especially some anti-epileptic drugs.

E13. Psychological, familial, sociological, geographical conditions that would limit compliance with study protocol requirements.

E14. Participation to another clinical trial that might interfere with the evaluation of the main criterion.

E15. Known hypersensitivity to the active substance or to any of the excipients of cabozantinib.

E16. Patient requiring tutorship or curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
The non progression rate in brain metastases at 6 months | At 6 months for each patient
  Tumor assessment in brain will be performed by cerebral MRI at baseline, 1.5 months, 3 months and 6 months. These cerebral MRI will be reviewed by central review according to the RANO-BM criteria.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 54 months
  Assessed using the National Cancer Institute - Common Terminology Criteria for Adverse Event (NCI-CTCAE) v5 grading scale, specific registration of neurological event during study duration.
Best response in brain metastases | Up to follow-up visit month 18 for each patient
  Evaluated according to RANDO-BM criteria.
Duration of response in brain | Up to 18 months for each patient
  From the date of inclusion to the date of first documented disease progression.
Progression-free survival | Up to 18 months for each patient
  Measured from the date of inclusion to the date of first documented disease progression or death from any cause.
Overall survival | Up to 54 months
  Measured from the date of inclusion to the date of death from any cause.
Response rate on the extracranial disease at 3 and 6 months | From baseline to 3 months and 6 months for each patients
  Defined as the poportion of patients with a complete or a partial response at 3 and 6 months, evaluated according to RECIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie NEGRIER, MD,PhD, Principal Investigator — Centre Leon Berard
Locations (12):
- France (12):
  - Institut de Cancérologie de l'Ouest-Site Paul Papin, Angers
  - CHU Besancon, Besançon
  - CHU Bordeaux, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Leon Berard, Lyon
  - Institut de Cancérologie de la Lorraine, Nancy
  - Hopital Européen Georges Pompidou, Paris
  - Institut de Cancérologie de l'Ouest-site René Gauducheau, Saint-Herblain
  - ICANS, Strasbourg
  - Hopital Foch, Suresnes
  - IUCT-Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif